CLINICAL TRIAL: NCT03328832
Title: Comparison of Combined Topical Tranexamic Acid With Floseal® With Intravenous Tranexamic Acid on Blood Loss in Total Knee Arthroplasty
Brief Title: Combined Topical Tranexamic Acid With Floseal® in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Jun-Wen, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201601271A0
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Thrombin-gelatin matrix; Floseal; Tranexamic Acid; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; Tranylcypromine; FloSeal Matrix; Rivaroxaban

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combined topical TXA and Floseal (Active Comparator): Floseal® was applied on potential bleeding sites before prosthesis implantation, and intraarticular application of topical tranexamic acid after capsule closure Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14.
  Interventions: Drug: Topical tranexamic acid; Drug: Floseal®; Drug: rivaroxaban (10mg)
- Topical TXA alone (Active Comparator): Intraarticular application of topical tranexamic acid after capsule closure Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14.
  Interventions: Drug: Topical tranexamic acid; Drug: rivaroxaban (10mg)

INTERVENTIONS:
Drug: Topical tranexamic acid — Intraarticular application of tranexamic acid 3g in 60 ml normal saline into knee joint after closure of the joint capsule
  Other Names: Topical transamine
Drug: Floseal® — Floseal® (Hemostatic matrix, 10ml, Baxter) was applied on potential bleeding sites: the femoral insertion of the posterior cruciate ligament, the lateral genicular artery after resection of the meniscus, the posterior capsule of the knee joint, the bony surfaces not covered by the implant as well as the pinholes (femur and tibia). The entire content of a 10 mL vial containing the active product (Floseal®) was used. The HM remained in place for 3 minutes and was then gently rinsed from the knee as recommended by the manufacturer (Baxter)
  Other Names: Thrombin-gelatin matrix
  Arms: Combined topical TXA and Floseal
Drug: rivaroxaban (10mg) — Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14.
  Other Names: Xarelto

SUMMARY:
Our purpose of this study therefore is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of combined topical application of these two hemostatic agents in different time during surgery and the safety compared with single topical application of TKA in a primary TKA procedure

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with considerable blood loss and increasing needs for allogenic blood transfusion. Tranexamic acid (TXA), an inhibitor of fibrinolysis, was reportedly effective reducing blood loss after standard TKA. Our previous experiences in minimally invasive (MIS) TKA showed that intraoperative infusion of TXA reduced 45% of postoperative blood loss and needs for transfusion from 20% to 4%. There were some reports demonstrating the cost-effectiveness of topical application of TXA in TKA patients.

Besides, thrombin-based hemostatic agents, Floseal®(Baxter, Deerfield, Illinois), have been widely used in surgical procedure. Some recent studies demonstrated that topical use of Floseal® in primary TKA can reduce hemoglobin decline and calculated total blood loss after TKA. But other studies showed Floseal® does not reduce blood loss in TKA procedures.

We believe the topical use of hemostatic agent in patients with high risk of thromboembolism can avoid its systematic effect and decrease its potential perioperative risk of thromboembolic complications (arterial thrombosis, myocardial infarction and pulmonary embolism). Recently, there were some reports demonstrating the cost-effectiveness of topical application of TXA in TKA patients. The blood saving effect of topical application of TXA in primary TKA was similar with systemic administration. The mean total blood loss of topical route of TXA inTKA patients was 940-1295 ml in different reports which was still high for patients with high thromboembolic risks. However, the efficacy and safety of topical use of TXA in TKA patients with history of thromboembolic disease is still unclear. A more effective regimen for bleeding prophylaxis afer primary TKA is necessary.

We believe that combined topical applications of two hemostatic agents of different mechanisms can bring a synergistic effect in blood saving and does not increase the risk of thromboembolic disease after TKA.

Our purpose of this study therefore is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of combined topical application of these two hemostatic agents in different time during surgery and the safety compared with single topical application of TKA in a primary TKA procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have advanced knee osteoarthritis are scheduled to undergo primary, unilateral elective total knee replacement surgery
2. Age > 50 years and < 90 years
3. Failure of medical treatment or rehabilitation.
4. Hemoglobin > 11g/dl,
5. No use of non-steroid anti-inflammatory agent one week before operation

Exclusion Criteria:

1. Preoperative Hemoglobin ≦11 g/dl
2. History of infection or intraarticular fracture of the affective knee
3. Renal function deficiency (GFR <30 ml/min/1.73m2)which is relative contraindicated for chemical venous thromboembolism
4. Elevated liver enzyme (AST/ALT level are more than twice normal range) , history of liver cirrhosis, impaired liver function(elevated total bilirubin level) and coagulopathy (including long-term use anticoagulant)
5. History of deep vein thrombosis, ischemic heart disease or stroke
6. Contraindications of tranexamic acid, floseal, or rivaroxaban
7. Allergy to tranexamic acid, floseal, rivaroxaban, or the excipients
8. History of heparin-induced thrombocytopenia (HIT)
9. Coagulopathy or bleeding tendency caused by organ dysfunction, such as cirrhosis, bone marrow suppression etc.
10. Patient who have active bleeding disorder, such as intracranial hemorrhage, upper GI bleeding, hematuria.
11. Patients with known allergies to materials of bovine origin

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Wen Wang, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets used and analyzed in the study are available on request to the corresponding author

REFERENCES:
- [Background] Bong MR, Patel V, Chang E, Issack PS, Hebert R, Di Cesare PE. Risks associated with blood transfusion after total knee arthroplasty. J Arthroplasty. 2004 Apr;19(3):281-7. doi: 10.1016/j.arth.2003.10.013. PMID 15067638
- [Background] Bierbaum BE, Callaghan JJ, Galante JO, Rubash HE, Tooms RE, Welch RB. An analysis of blood management in patients having a total hip or knee arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):2-10. doi: 10.2106/00004623-199901000-00002. PMID 9973048
- [Background] Goodnough LT, Verbrugge D, Marcus RE. The relationship between hematocrit, blood lost, and blood transfused in total knee replacement. Implications for postoperative blood salvage and reinfusion. Am J Knee Surg. 1995 Summer;8(3):83-7. PMID 7552610
- [Background] Tanaka N, Sakahashi H, Sato E, Hirose K, Ishima T, Ishii S. Timing of the administration of tranexamic acid for maximum reduction in blood loss in arthroplasty of the knee. J Bone Joint Surg Br. 2001 Jul;83(5):702-5. doi: 10.1302/0301-620x.83b5.11745. PMID 11476309
- [Background] Alvarez JC, Santiveri FX, Ramos I, Vela E, Puig L, Escolano F. Tranexamic acid reduces blood transfusion in total knee arthroplasty even when a blood conservation program is applied. Transfusion. 2008 Mar;48(3):519-25. doi: 10.1111/j.1537-2995.2007.01564.x. Epub 2007 Dec 7. PMID 18067499
- [Background] Petaja J, Myllynen P, Myllyla G, Vahtera E. Fibrinolysis after application of a pneumatic tourniquet. Acta Chir Scand. 1987 Nov-Dec;153(11-12):647-51. PMID 3124428
- [Background] Kambayashi J, Sakon M, Yokota M, Shiba E, Kawasaki T, Mori T. Activation of coagulation and fibrinolysis during surgery, analyzed by molecular markers. Thromb Res. 1990 Oct 15;60(2):157-67. doi: 10.1016/0049-3848(90)90294-m. PMID 2149215
- [Background] Hiippala S, Strid L, Wennerstrand M, Arvela V, Mantyla S, Ylinen J, Niemela H. Tranexamic acid (Cyklokapron) reduces perioperative blood loss associated with total knee arthroplasty. Br J Anaesth. 1995 May;74(5):534-7. doi: 10.1093/bja/74.5.534. PMID 7772427
- [Background] Benoni G, Fredin H. Fibrinolytic inhibition with tranexamic acid reduces blood loss and blood transfusion after knee arthroplasty: a prospective, randomised, double-blind study of 86 patients. J Bone Joint Surg Br. 1996 May;78(3):434-40. PMID 8636182
- [Background] Ido K, Neo M, Asada Y, Kondo K, Morita T, Sakamoto T, Hayashi R, Kuriyama S. Reduction of blood loss using tranexamic acid in total knee and hip arthroplasties. Arch Orthop Trauma Surg. 2000;120(9):518-20. doi: 10.1007/s004029900132. PMID 11011672
- [Background] Lin PC, Hsu CH, Chen WS, Wang JW. Does tranexamic acid save blood in minimally invasive total knee arthroplasty? Clin Orthop Relat Res. 2011 Jul;469(7):1995-2002. doi: 10.1007/s11999-011-1789-y. Epub 2011 Feb 1. PMID 21286886
- [Background] Graham ID, Alvarez G, Tetroe J, McAuley L, Laupacis A. Factors influencing the adoption of blood alternatives to minimize allogeneic transfusion: the perspective of eight Ontario hospitals. Can J Surg. 2002 Apr;45(2):132-40. PMID 11939657
- [Background] Nishihara S, Hamada M. Does tranexamic acid alter the risk of thromboembolism after total hip arthroplasty in the absence of routine chemical thromboprophylaxis? Bone Joint J. 2015 Apr;97-B(4):458-62. doi: 10.1302/0301-620X.97B4.34656. PMID 25820882
- [Background] Xie J, Ma J, Kang P, Zhou Z, Shen B, Yang J, Pei F. Does tranexamic acid alter the risk of thromboembolism following primary total knee arthroplasty with sequential earlier anticoagulation? A large, single center, prospective cohort study of consecutive cases. Thromb Res. 2015 Aug;136(2):234-8. doi: 10.1016/j.thromres.2015.05.014. Epub 2015 May 21. PMID 26026635
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PMID 23541868
- [Background] Chimento GF, Huff T, Ochsner JL Jr, Meyer M, Brandner L, Babin S. An evaluation of the use of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):74-7. doi: 10.1016/j.arth.2013.06.037. PMID 24034510
- [Background] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406
- [Background] Georgiadis AG, Muh SJ, Silverton CD, Weir RM, Laker MW. A prospective double-blind placebo controlled trial of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):78-82. doi: 10.1016/j.arth.2013.03.038. Epub 2013 Jul 29. PMID 23906869
- [Background] Gazzeri R, Galarza M, Alfier A. Safety biocompatibility of gelatin hemostatic matrix (Floseal and Surgiflo) in neurosurgical procedures. Surg Technol Int. 2012 Dec;22:49-54. PMID 22915500
- [Background] Clapp M, Huang JC. Use of FloSeal Sealant in the Surgical Management of Tubal Ectopic Pregnancy. Case Rep Obstet Gynecol. 2013;2013:906825. doi: 10.1155/2013/906825. Epub 2013 May 29. PMID 23819082
- [Background] Testini M, Marzaioli R, Lissidini G, Lippolis A, Logoluso F, Gurrado A, Lardo D, Poli E, Piccinni G. The effectiveness of FloSeal matrix hemostatic agent in thyroid surgery: a prospective, randomized, control study. Langenbecks Arch Surg. 2009 Sep;394(5):837-42. doi: 10.1007/s00423-009-0497-5. Epub 2009 May 7. PMID 19421770
- [Background] Di Francesco A, Flamini S, Fiori F, Mastri F. Hemostatic matrix effects on blood loss after total knee arthroplasty: A randomized controlled trial. Indian J Orthop. 2013 Sep;47(5):474-81. doi: 10.4103/0019-5413.118203. PMID 24133307
- [Background] Suarez JC, Slotkin EM, Alvarez AM, Szubski CR, Barsoum WK, Patel PD. Prospective, randomized trial to evaluate efficacy of a thrombin-based hemostatic agent in total knee arthroplasty. J Arthroplasty. 2014 Oct;29(10):1950-5. doi: 10.1016/j.arth.2014.05.025. Epub 2014 Jun 5. PMID 25015756
- [Background] Kim HJ, Fraser MR, Kahn B, Lyman S, Figgie MP. The efficacy of a thrombin-based hemostatic agent in unilateral total knee arthroplasty: a randomized controlled trial. J Bone Joint Surg Am. 2012 Jul 3;94(13):1160-5. doi: 10.2106/JBJS.K.00531. PMID 22623075
- [Background] Helito CP, Gobbi RG, Castrillon LM, Hinkel BB, Pecora JR, Camanho GL. Comparison of Floseal(r) and electrocautery in hemostasis after total knee arthroplasty. Acta Ortop Bras. 2013;21(6):320-2. doi: 10.1590/S1413-78522013000600004. PMID 24453689
- [Background] Comadoll JL, Comadoll S, Hutchcraft A, Krishnan S, Farrell K, Kreuwel HT, Bechter M. Comparison of hemostatic matrix and standard hemostasis in patients undergoing primary TKA. Orthopedics. 2012 Jun;35(6):e785-93. doi: 10.3928/01477447-20120525-14. PMID 22691647
- [Background] Bae KC, Cho CH, Lee KJ, Son ES, Lee SW, Lee SJ, Lim KH. Efficacy of intra-articular injection of thrombin-based hemostatic agent in the control of bleeding after primary total knee arthroplasty. Knee Surg Relat Res. 2014 Dec;26(4):236-40. doi: 10.5792/ksrr.2014.26.4.236. Epub 2014 Dec 2. PMID 25505706
- [Background] Schwab PE, Thienpont E. Use of a haemostatic matrix does not reduce blood loss in minimally invasive total knee arthroplasty. Blood Transfus. 2015 Jul;13(3):435-41. doi: 10.2450/2015.0199-14. Epub 2015 Jan 26. PMID 25761324
- [Background] Schwab PE, Thienpont E. Use of a haemostatic matrix (Floseal(R)) does not reduce blood loss in minimally invasive total knee arthroplasty performed under continued aspirin. Blood Transfus. 2016 Mar;14(2):134-9. doi: 10.2450/2015.0023-15. Epub 2015 May 29. PMID 26057492
- [Background] Lin SY, Chen CH, Fu YC, Huang PJ, Chang JK, Huang HT. The efficacy of combined use of intraarticular and intravenous tranexamic acid on reducing blood loss and transfusion rate in total knee arthroplasty. J Arthroplasty. 2015 May;30(5):776-80. doi: 10.1016/j.arth.2014.12.001. Epub 2014 Dec 5. PMID 25534864

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2017 and September 2018, a consecutive series of 125 patients who underwent unilateral TKA were assessed in terms of their eligibility for inclusion for this study. 35 patients were excluded based on the exclusion criteria, eight patients did not withhold antiplatelet drugs or anticoagulants 7 days before surgery, and 12 other patients declined to participate in the study. Total 70 patients were enrolled and randomly assigned into 2 groups
Period: Overall Study
Arm/Group | Combined Topical TXA and Floseal | Topical TXA Alone
Started | 35 | 35
Completed | 35 | 34
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Topical TXA and Floseal | Topical TXA Alone | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.26 (5.88) | 67.47 (4.00) | 68.38 (4.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 34 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 35 | 34 | 69
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.69 (3.77) | 27.44 (4.44) | 28.07 (4.11)
Preop Hb [Mean (Standard Deviation); unit: g/dL] | 13.79 (1.39) | 13.39 (0.85) | 13.61 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss After Operation
Description: Total blood loss was calculated according to Nadler et al., which used maximum postoperative reduction of the Hb level adjust for weight and height of the patient. The formula is as follows, Total blood loss = (Total blood volume x [change in Hb level / preoperative Hb level])x1000+volume transfused
Time Frame: From the operation to the postoperative day 3 or 4
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Combined Topical TXA and Floseal | Topical TXA Alone
Number analyzed (Participants) | 35 | 34
ml | 678 (203) | 733 (217)
Statistical Analysis 1: Comparison: Combined Topical TXA and Floseal vs Topical TXA Alone; Test type: Equivalence — equivalence means p value > 0.05; p = 0.276, t-test, 2 sided

2. Secondary Outcome: Blood Transfusion Rate
Description: We will record the event of blood transfusion, and calculate the incidence of transfusion
Time Frame: From the operation to the postoperative day 3 or 4
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Topical TXA and Floseal | Topical TXA Alone
Number analyzed (Participants) | 35 | 34
Participants | 1 | 0
Statistical Analysis 1: Comparison: Combined Topical TXA and Floseal vs Topical TXA Alone; Test type: Equivalence — equivalence means p value > 0.05; p = 1, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Incidence of Thrombosis Events
Description: The composite of any venous thromoembolism events, ischemic heart attacks, cerebrovascular accidents
Time Frame: within 30 days of the operation
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Topical TXA and Floseal | Topical TXA Alone
Number analyzed (Participants) | 35 | 34
Participants | 0 | 0
Statistical Analysis 1: Comparison: Combined Topical TXA and Floseal vs Topical TXA Alone; Test type: Equivalence — Equivalence means p value > 0.05; p = 1, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Combined Topical TXA and Floseal | Topical TXA Alone
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 17/35 | 15/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Topical TXA and Floseal (N=35) | Topical TXA Alone (N=34)
Ecchymosis (Surgical and medical procedures) | 17 (17) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03328832/Prot_SAP_000.pdf